CLINICAL TRIAL: NCT01330056
Title: A Prospective Randomized Controlled Trial of Functional Organ Preservation Surgery vs. Chemoradiotherapy for Head and Neck Squamous Cell Carcinoma
Brief Title: Functional Organ Preservation Surgery
Acronym: FOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Lyel Roh, MD, PhD, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010-001
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-07

CONDITIONS: Organ Preservation
Keywords: Laryngeal and pharyngeal preservation, survivals
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FOPS (Active Comparator): * Functional organ preservation surgery (FOPS) group as a first-line treatment modality
  * Postoperative RT or CRT may be included for the patients of this group
  Interventions: Procedure: FOPS
- CRT (Active Comparator): * Concurrent chemoradiotherapy or radiotherapy group as a first-line treatment modality
  * Salvage surgery may be applied for the patients for persistent or recurrent cancers after CRT or RT
  Interventions: Radiation: CRT

INTERVENTIONS:
Procedure: FOPS — * Functional organ preservation (FOPS) as a first-line treatment modality
  * Postoperative RT or CRT may be included for the patients of this group.
  Arms: FOPS
Radiation: CRT — * Concurrent chemoradiotherapy as a first-line treatment modality
  * Salvage surgery may be applied for the patients with persistent or recurrent cancers after RT or CRT
  Arms: CRT

SUMMARY:
This is a prospective randomized controlled trial comparing functional organ preservation surgery (FOPS) vs. radiotherapy or chemoradiotherapy as the first treatment modality for patients with head an neck squamous cell carcinoma arising in the oropharynx, larynx and hypopharynx. This study has a hypothesis that the FOPS is an effective treatment strategy to preserve the organ function without compromising oncologic safety and survival.

DETAILED DESCRIPTION:
This prospective study compare the following items between two groups:

* Functional outcomes: laryngeal, pharyngeal, and quality of life
* Oncological outcomes: survivals, locoregional controls
* Combined imaging and molecular biomarkers with follow-up data

The functional organ preservation surgery (FOPS) is defined as a surgery preserving the laryngeal or pharyngeal function regardless of open or transoral route. The FOPS may include:

* Radical tonsillectomy or other oropharyngeal resection
* Partial laryngectomy or pharyngectomy
* Transoral laser microresection
* Transoral robotic surgery (TORS)
* Reconstructive surgery may be combined with primary resection
* Neck dissection may be indicated in some patients
* Postoperative radiotherapy or chemoradiotherapy may be indicated in some patients according to their pathologic reports.

The standard concurrent chemoradiotherapy (CRT) is generally used but radiotherapy (RT) alone may be indicated for some patients under tumor-board discussion. The salvage surgery may be indicated for patients with residual or recurrent diseases after CRT or RT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinomas arising in the oropharynx, larynx, or hypopharynx
* Resectable tumors without distant metastases
* age range: 18-80 years
* Pretreatment Karnofsky performance scale > or 70%
* Operable patients
* No significant loss of pretreatment larynx and pharyngeal functions

Exclusion Criteria:

* Patients with a present or previous history of other cancers except benign tumors, premalignant lesions, carcinoma-in-situ (at some organ sites), well-differentiated thyroid carcinoma and low-grade salivary gland cancers (from tumor-board decision whether the tumors significantly affect the survival outcomes)
* Other organ-site cancers
* Low-performance status or non-operable patients
* Non-resectable or distant-metastatic tumors
* Extensive primary or neck nodal diseases
* Significant pretreament loss of laryngeal or pharyngeal functions
* cT1N0 glottic carcinomas

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Actual)
Dates: Start 2010-09; Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Organ preservation rate | 2 years
  The larynge and pharyngeal functions are compared between two groups. The time frame may be extended to 5 years.

SECONDARY OUTCOMES:
Survival rate | 2 years
  The time frame may be extended to 5 years.
Locoregional control rate | 2 years
  The time frame may be extended to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Lyel Roh, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea